CLINICAL TRIAL: NCT05212753
Title: The Effect of Sleep Hygiene, Breathing and Stabilization Exercises on Pain, Sleep Quality and Anxiety Level in Patients With Chronic Non-Specific Low Back Pain
Brief Title: The Effect of Breathing Exercise and Stabilization Exercise With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Samed Gulyilmaz, Principal Investigator, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/031
Record Dates: First submitted 2022-01-16; First posted 2022-01-28 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2022-01

CONDITIONS: Low Back Pain; Sleep Hygiene; Anxiety
Keywords: Nonspecific Chronic Low Back Pain; Sleep Quality; Breathing Exercises
MeSH Terms: conditions — Low Back Pain; Sleep Hygiene; Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Physical Therapy Group (Active Comparator): The conventional physical therapy group will receive Transcutaneous Electrical Nerve Stimulation (TENS) and hot pack application.
  Interventions: Device: Conventional physical therapy
- Stabilization Group (Active Comparator): The stabilization group will receive lumbar stabilization exercises and the conventional physical therapy program. That program includes lumbar stabilization exercises including activation of the transverses abdominals (TA) and multifidi muscles.
  Interventions: Device: Conventional physical therapy; Other: Lumbar stabilization exercises
- Breathing Exercise Group (Active Comparator): The breathing exercise group will receive breathing exercises including sleep hygiene, and the stabilization group program. Breathing exercises include diaphragmatic breathing and pursed-lip.
  Interventions: Device: Conventional physical therapy; Other: Lumbar stabilization exercises; Other: Breathing exercises

INTERVENTIONS:
Device: Conventional physical therapy — Hot packs or hot water bags are superficial warming agents that will be used to heat muscle tissue, reduce muscle spasms and pain sensation. TENS is a pain reliever application.
Other: Lumbar stabilization exercises — Training about the concepts of stabilization and abdominal bracing is given before starting the study. The motor control tests for local muscles transversus abdominus and multifidi are performed after the training. The abdominal bracing test is performed in the quadruped position, in prone, and in hook lying position with the patient's spine supine with hips and knees flexed and knees in contact with the surface. The second stage consists of closed-chain segmental control exercises. It is a series of weight-bearing exercises are performed on stable and unstable surfaces. The last stage of the stabilization program is an open kinetic chain exercise to promote distal stability.
  Arms: Breathing Exercise Group; Stabilization Group
Other: Breathing exercises — Breathing exercises consist of the techniques of diaphragmatic and pursed-lip breathing. During diaphragmatic breathing, attention is focused on the correct abdominal breathing. The pursed-lip breathing is one step further to the diaphragmatic breathing and a technique designed to have control time and volume over-breathing. This intervention also includes Sleep Hygiene education to the subjects,
  Arms: Breathing Exercise Group

SUMMARY:
The aim of this study is to compare the effect of sleep hygiene, breathing exercises, and stabilization exercises on pain, sleep quality, and anxiety level in patients with non-specific chronic low back pain.

DETAILED DESCRIPTION:
Addressing sleep problems in patients with chronic non-specific low back pain (LBP) can reduce chronic pain, the risk of developing depressive illness and improve pain-related quality of life.

Sleep is a concept that has physiological, psychological, and social dimensions. Sleep is one of the essential and indispensable daily life activities that affect individuals' quality of life and well-being. Decreasing pain is expected and likely to improve sleep quality. Still, it is unknown what will happen due to improving sleep quality to resolve the pain of unknown origin.

Education about sleep hygiene with physiotherapy has not been assessed before on individuals with nonspecific LBP. Since this training will require a lifestyle change, individuals should be warned not once but several times in a certain time, and this training should be reinforced. This will be an advantage for the patients receiving physiotherapy, and their therapists will support them in applying this training during the physiotherapy sessions.

In our study, individuals with nonspecific chronic low back pain will be divided into three groups using the blinding method as part of a randomized controlled trial.

The first group, as the conventional physical therapy group, will receive a hot pack and TENS only.

The second group, as the stabilization group, will receive lumbar stabilization exercises and the conventional physical therapy program.

The third group, as the breathing exercise group, will receive breathing exercises, including sleep hygiene and stabilization group program.

ELIGIBILITY:
Inclusion Criteria:

* individuals between the ages of 18-65
* Having low back pain for at least the last 3 months
* Pain at 4 out of 10 according to VAS (Visual Analogue Scale)

Exclusion Criteria:

* Radiculopathies
* Body mass index > 35
* Neurological, orthopedic, or cardiopulmonary diseases that will contraindicate exercise
* Treatment for pain in the last 3 months who have received
* individuals who can't cooperate and those who have problems adapting to exercises

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pain at 3 weeks and 8 weeks | Baseline, 3 weeks, 8 weeks
  Visual Analogue Scale will be used where patients will be asked to rate their pain on a scale from 0 to 10 with 0 indicating no pain and 10 the maximum worst pain, at the baseline and the end of 3 weeks intervention and at the end 8 weeks from baseline.
Change from Baseline in Form of Pain at 3 weeks and 8 weeks | Baseline, 3 weeks, 8 weeks
  Form of Pain will be assessed with the Mcgill Melzack Pain Questionnaire. The questionnaire consists of four parts. In the first part, the individual marks the place where they feel pain on a representative body picture and indicates with the letters "D" if the pain is deep, "S" if it is on the body surface, and "D-S" if it is both deep and superficial. In the second part, there are 20 statements that examine pain from various aspects. The individual is asked to choose the word group that fits their pain and to marks only one word in the selected group that fits their pain. In the third part, there are questions about the relationship between time and pain. In the fourth part, five word-groups ranging from "mild to unbearable" pain are defined to determine the severity of pain.
Change from Baseline in Sleep Quality at 3 weeks and 8 weeks | Baseline, 3 weeks, 8 weeks
  Sleep quality will be assessed with the Pittsburgh Sleep Quality Index (PSQI). PSQI is a 19-item self-report questionnaire that measures subjective sleep quality over the previous month. The individual 19 items in the PSQI are aggregated into seven components that assess various aspects of sleep, and the sum of these seven components yields a score that distinguishes between "good" and "bad" sleepers.
Change from Baseline in Anxiety at 3 weeks and 8 weeks | Baseline, 3 weeks, 8 weeks
  Anxiety will be assessed with the Spielberger State-Trait Anxiety Inventory. It consists of two separate scales, each with 20 questions, assessing the levels of state anxiety and trait anxiety. The score that can be obtained from both scales is a minimum of 20 and a maximum of 80. If the score from the scale is high, the person's anxiety is high.
Change from Baseline in Fatigue at 3 weeks and 8 weeks | Baseline, 3 weeks, 8 weeks
  Fatigue will be assessed with the Fatigue Severity Scale.
  This scale consists of 9 items in total. Individuals give points from 1 to 7 for each item. If the average score is greater than 6.1, it is concluded as chronic fatigue.

SECONDARY OUTCOMES:
Obstructive Sleep Apnea Risk Screening İn İndividuals With Chronic Non-Specific Low Back Pain | Baseline
  Stop-Bang Survey, used as a screening tool for obstructive sleep apnea (OSAS), is a questionnaire consisting of 8-item yes/no responses with a score for each positive answer.
  Moderate risk of OSAS: yes to 3-4 questions, and high risk of OSAS: yes to 5-8 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Aysenur Tuncer, PhD, Study Director — Hasan Kalyoncu University
Locations (1):
- İslahiye İlçe Hast., Gaziantep, Turkey (Türkiye)